CLINICAL TRIAL: NCT04485182
Title: Underwater Jet Massage Therapy for Chronic Low Back Pain
Status: Terminated | Type: Observational
Why Stopped: Due to the COVID pandemia the tubes of the treatments baths went wrong.
Sponsor: Polyclinic of the Hospitaller Brothers of St. John of God, Budapest (Other)
Responsible Party: Principal Investigator, Tamas Gati, 1027 Budapest Árpád fejedelem út 7., Polyclinic of the Hospitaller Brothers of St. John of God, Budapest
Other Study IDs: PolyclinicHBSJG
Record Dates: First submitted 2020-04-12; First posted 2020-07-24 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain
Keywords: hydrotherapy, massage
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First: Patients receiving Transcutaneous Electrical Nerve Stimulation + underwater massage + spine gymnastics +
  Interventions: Other: Underwater jet massage (Tangentor)
- controll group: Patients receiving Transcutaneous Electrical Nerve Stimulation + spine gymnastics

INTERVENTIONS:
Other: Underwater jet massage (Tangentor) — Underwater jet massage (Tangentor) would be performed in a tub developed for this purpose, where the water temperature: 33-35 ° C. The treatments lasting from 15 atm and 15 cm for 15 minutes.
  They take a minimum of 10 treatments for approx. under 2 weeks.
  Groups: First

SUMMARY:
Underwater massage is the more modern variety of massages otherwise known as tangentor, where the temperature of the water of the treatment tub and the mechanical effect of the water jet is utilised. It is typical of chronic low back pain that, after the first painful episode, is repeated at 44-78% of patients.

Our goals are the followings:

1. Is the beneficial effect of a Underwater massage therapy addition to a complex physiotherapy comparable to a control group with respect to clinical parameters?
2. How much does the quality of life change in an initial state and how much is it in comparison with the control group?

DETAILED DESCRIPTION:
Informed consent was obtained from all participants. We use two groups to investigate the effects of the tangentor on the low back pain.

The patients presenting at the rheumatology inpatient clinics were enrolled without into the treatment and control groups.

Patients receiving Transcutaneous Electrical Nerve Stimulation + underwater massage + spine gymnastics

In the controll group the Patients receiving Transcutaneous Electrical Nerve Stimulation + spine gymnastics

Underwater jet massage (Tangentor) would be performed in a tub developed for this purpose, where the water temperature: 33-35 ° C. The treatments lasting from 15 atm and 15 cm for 15 minutes.

The water temperature is precisely measured by a built-in thermometer. Pressure is controlled by a manometer.

They take a minimum of 10 treatments for approx. under 2 weeks.

The back massage position is, that the patient lying on their side, hip and knees are slightly bent and the head and neck rest on a support.

After the massage the client should rest for about 30minutes.

Patients participated in two visits, for the first time before the study, right after the therapy treatments.

During the study, all participants received the usual or necessary medications. On a Visual Analogue Scale (VAS) patients indicated degree of pain on a scale from 0 to 100 mm for the past week. VAS scores were expressed in millimetres (zero point-no pain; endpoint-intolerable pain). Patients recorded on the VAS scale the level of low back pain at rest as well as during activity. Functional disability was assessed by using the Oswestry Disability Index (ODI).

Furthermore, there was a questionnaire on the quality of life, known as the EuroQol Five Dimensions Questionnaire (EQ-5D-5L).

ELIGIBILITY:
Inclusion Criteria:

* at least 12 weeks of non-specific lymphatic pain,the pain sensitivity of the paravertebral muscle and the painful movement of the lumbar spine can be observed, which can be characterized by segmental motion, segmental instability or other reasons.
* radiographically confirmed spondylosis, discopathy, and spondylarthrosis within one year.
* back pain at least 30mm (100mm visualis analogue scale).
* patient consent form signed before the start of test

Exclusion Criteria:

* patients could not received systemic or locally administered steroid therapy, physiotherapy or they get balneotherapy in the last 2 months
* The exclusion criteria included:
* previous lumbar spine surgery,
* progressive neurologic loss,
* pregnancy,
* umbilical- , inguinal hernia,
* malignities,
* infectious diseases,
* inflammatory pathologies,
* severe pulmonary and cardiovascular diseases,
* uncontrolled hypertension,
* mental disorders,
* incontinence,
* Acute lower back pain; Organic neurological symptoms associated with the lower back;
* pain in the background of osteoporosis or other causes of vertebral compression is likely; malignity in the background;
* Lack of complience,
* Pain due to inflammatory spinal disease;
* spondylolisthesis (which is not greater than 25% of vertebral skeleton compared to adjacent vertebrae)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Enrollment criteria were as follows: outpatients aged 18-85 with non-specific low back pain that persists for at least 12 weeks, showing degenerative symptoms and suffering from moderately reduced mobility. Patient's pain intensity during activity should have been minimum 30mm on Visual Analogue Scale (0-100 mm VAS).
  Written information on the methodology and process they would be undergoing was provided to each participant, and an informed consent form was subsequently signed before the study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Tangentor | 2 years
  Investigate the beneficial effect of a Underwater massage therapy addition to a complex physiotherapy comparable to a control group with respect to clinical parameters on a Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Tangentor | 2 years
  How much does the quality of life change in an initial state and how much is it in comparison with the control group on the EuroQol Five Dimensions Questionnaire (EQ-5D-5L).

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinic of the Hospitaller Brothers of St. John of God,, Budapest, Árpád Fejedelem Útja 7, Hungary